CLINICAL TRIAL: NCT04390971
Title: A Multi-center, Open Label Study to Evaluate the Safety and Efficacy of ET-01 Transplantation in Subjects With Transfusion Dependent β-Thalassemia
Brief Title: Safety and Efficacy Evaluation of ET-01 Transplantation in Subjects With Transfusion Dependent β-Thalassaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: EdiGene Inc. (Industry); The Affiliated Hospital Of Guizhou Medical University (Other); Zunyi Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC2019004
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2023-11

CONDITIONS: Transfusion Dependent Beta-Thalassaemia
Keywords: Beta-Thalassaemia; Hematopoietic Stem-Cell Transplantation
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ET-01 (Experimental): BCL11A Enhancer modified Autologous Hematopoietic Stem Cells.
  Interventions: Biological: ET-01

INTERVENTIONS:
Biological: ET-01 — Recruited participants will receive ET-01 IV infusion after conditioning.

SUMMARY:
This is an open label, multi-center study to evaluate the safety and Efficacy of ET-01 Transplantation in subjects with Transfusion Dependent β-Thalassaemia.

DETAILED DESCRIPTION:
After the proper subject is recruited, subject will go through steps generally as stem cell mobilization, apheresis, conditioning and ET-01 infusion to complete therapy. Two years follow-up will be carried out post-transplantation and related data will be collected. Subjects who have been treated by ET-01 will be asked to participate in a long-term follow up study. Monitoring the long-term efficacy and safety up to 15 years after ET-01 transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or subject's legal personal representative fully understand and voluntarily sign informed consent forms;
* 6~35 years old, all gender;
* Diagnosis of transfusion dependent β-thalassemia (β-TDT) as defined by protocol;
* Eligible for autologous stem cell transplant;
* Eligible for autologous stem cell transplant;
* Organs in good function.
* Other protocol defined inclusion criteria may apply.

Exclusion Criteria:

* Subjects with associated α-thalassemia;
* Active bacterial, virus, fungal or parasitic infection, including HIV infection, HbsAg and HBV DNA positive, HCV DNA positive, or Treponema Pallidum infection;
* HLA identical sibling or unrelated donors are available;
* Prior allo-HSCT or gene therapy.
* Other protocol defined exclusion criteria may apply.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs & SAEs identified according to NCI CTCAE 5.0. | From ET-01 infusion to 104 weeks post-transplant
All-cause mortality | From signing of informed consent to 104 weeks post-transplant
Incidence of transplant-related mortality | Within 100 days post-transplant
Proportion of subjects with engraftment | Up to 42 days post-transplant

SECONDARY OUTCOMES:
Change of total hemoglobin from baseline | Within 104 weeks post-transplant
Change of HbF from baseline | Within 104 weeks post-transplant
Change of proportion of HbF/Hb | Within 104 weeks post-transplant
Change of frequency of packed RBC transfusions | From 6 months before recruitment to 104 weeks post-transplant
Change of volume of packed RBC transfusions | From 6 months before recruitment to 104 weeks post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (3):
- China (3):
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No